CLINICAL TRIAL: NCT07337265
Title: Effect of Oral Royal Jelly Supplementation on Sperm DNA Fragmentation Index and Pregnancy in Couples With Unexplained Infertility: A Prospective, Randomized, Double-Blind, Placebo-Controlled Clinical Study
Brief Title: Royal Jelly Supplementation in Unexplained Male Infertility
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Ali Ihsan Memmi, medical doctor, Medipol University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 123123123123
Record Dates: First submitted 2026-01-01; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Unexplained Infertility; Male Infertility; Sperm DNA Fragmentation
Keywords: royal jelly; unexplained male infertility; sperm dna fragmentation
MeSH Terms: conditions — Infertility, Male

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Royal Jelly (Experimental): Participants will receive 750 mg of Lyophilized Royal Jelly capsules daily for 3 months (90 days).
  Interventions: Dietary Supplement: Lyophilized Royal Jelly
- Placebo Group (Placebo Comparator): Participants will receive inert capsules identical in appearance and taste to the experimental drug daily for 3 months (90 days).
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Lyophilized Royal Jelly — Participants will receive 750 mg of Lyophilized Royal Jelly capsules daily for 3 months (90 days).
  Arms: Royal Jelly
Other: Placebo — Participants will receive inert capsules identical in appearance and taste to the experimental drug daily for 3 months (90 days)
  Arms: Placebo Group

SUMMARY:
This randomized, double-blind, placebo-controlled clinical trial investigates the effects of oral Royal Jelly supplementation on sperm DNA fragmentation and pregnancy rates in couples with unexplained infertility. While routine semen analysis appears normal (normozoospermia) in these patients, underlying Sperm DNA Fragmentation (SDF) and oxidative stress are believed to contribute to reproductive failure.

Participants will be randomized to receive either 750 mg of lyophilized Royal Jelly or a placebo daily for a period of 3 months (90 days). The study aims to evaluate whether the antioxidant properties of Royal Jelly can improve sperm chromatin integrity, reduce oxidative stress markers, and increase spontaneous pregnancy rates compared to the control group

DETAILED DESCRIPTION:
Infertility is a global health issue affecting approximately 15% of couples. "Unexplained Infertility" constitutes about 15-30% of these cases, where standard diagnostic tests (semen analysis, ovulation tests, and tubal patency) appear normal. Major factors contributing to the etiology of unexplained infertility include Sperm DNA Fragmentation (SDF) and Seminal Oxidative Stress (OS), which are not detected in routine spermiograms but can impair fertilization.

The European Association of Urology (EAU) guidelines suggest SDF testing in unexplained infertility cases, as high SDF rates reduce natural pregnancy chances and the success of assisted reproductive techniques. Royal Jelly, rich in 10-hydroxy-2-decenoic acid (10-HDA) and flavonoids, possesses potent antioxidant properties. While previous studies have shown that Royal Jelly improves sperm parameters, its efficacy specifically on DNA integrity in normozoospermic men with unexplained infertility remains unknown.

This prospective, randomized, double-blind, placebo-controlled study aims to investigate the protective effect of oral Royal Jelly supplementation on sperm DNA integrity and spontaneous pregnancy rates in men with unexplained infertility.

ELIGIBILITY:
Inclusion Criteria:

* Men aged 18-45 years. History of infertility for at least 1 year despite unprotected intercourse.

Diagnosis of unexplained infertility with Normozoospermia according to WHO 2021 (6th Ed.) criteria:

Concentration ≥ 16 million/mL Total Motility ≥ 42% Progressive Motility ≥ 30% Normal Morphology (Kruger) ≥ 4% Female partner with normal gynecological evaluation (regular ovulation, normal ovarian reserve, and proven tubal patency via HSG).

Normal serum hormone levels (Testosterone, FSH, LH)

Exclusion Criteria:

* Any abnormality in spermiogram (Oligo-, Asteno-, or Teratozoospermia). Presence of clinical varicocele. Leukocytospermia (>1 million/mL) or active infection. History of smoking (>5 cigarettes/day) or BMI > 30 kg/m². Use of any antioxidant supplementation within the last 3 months.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 80 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Change in Sperm DNA Fragmentation Index (SDF) | Baseline (Day 0) and Post-treatment (Day 90)
  DNA damage will be assessed using the HaloSperm to determine the percentage of spermatozoa with fragmented DNA
Spontaneous Pregnancy Rate | Up to 3 months (90 days)
  Number of couples achieving spontaneous pregnancy during the study period.

SECONDARY OUTCOMES:
Serum Hormonal Profile | Baseline (Day 0) and Post-treatment (Day 90)
  Measurement of serum Total Testosterone, FSH, and LH levels.
Seminal Oxidative Stress Markers (TAS/TOS/OSI) | Baseline (Day 0) and Post-treatment (Day 90)
  Evaluation of Total Antioxidant Status (TAS), Total Oxidant Status (TOS), and Oxidative Stress Index (OSI) using spectrophotometric analysis.
Sperm Chromatin Integrity | Baseline (Day 0) and Post-treatment (Day 90)
  Assessment of chromatin integrity using Toluidine Blue staining.
Immunohistochemical Analysis (Exploratory) | Baseline (Day 0) and Post-treatment (Day 90)
  Evaluation of Mapk erk 1/2, Pten, and Mtor antibody expression in sperm samples.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Amirshahi T, Najafi G, Nejati V. Protective effect of royal jelly on fertility and biochemical parameters in bleomycin-induced male rats. Iran J Reprod Med. 2014 Mar;12(3):209-16. PMID 24799882
- [Result] Tharakan T, Bettocchi C, Carvalho J, Corona G, Jones TH, Kadioglu A, Salamanca JIM, Serefoglu EC, Verze P, Salonia A, Minhas S; EAU Working Panel on Male Sexual Reproductive Health. European Association of Urology Guidelines Panel on Male Sexual and Reproductive Health: A Clinical Consultation Guide on the Indications for Performing Sperm DNA Fragmentation Testing in Men with Infertility and Testicular Sperm Extraction in Nonazoospermic Men. Eur Urol Focus. 2022 Jan;8(1):339-350. doi: 10.1016/j.euf.2020.12.017. Epub 2021 Jan 6. PMID 33422457
- [Result] Agarwal A, Parekh N, Panner Selvam MK, Henkel R, Shah R, Homa ST, Ramasamy R, Ko E, Tremellen K, Esteves S, Majzoub A, Alvarez JG, Gardner DK, Jayasena CN, Ramsay JW, Cho CL, Saleh R, Sakkas D, Hotaling JM, Lundy SD, Vij S, Marmar J, Gosalvez J, Sabanegh E, Park HJ, Zini A, Kavoussi P, Micic S, Smith R, Busetto GM, Bakircioglu ME, Haidl G, Balercia G, Puchalt NG, Ben-Khalifa M, Tadros N, Kirkman-Browne J, Moskovtsev S, Huang X, Borges E, Franken D, Bar-Chama N, Morimoto Y, Tomita K, Srini VS, Ombelet W, Baldi E, Muratori M, Yumura Y, La Vignera S, Kosgi R, Martinez MP, Evenson DP, Zylbersztejn DS, Roque M, Cocuzza M, Vieira M, Ben-Meir A, Orvieto R, Levitas E, Wiser A, Arafa M, Malhotra V, Parekattil SJ, Elbardisi H, Carvalho L, Dada R, Sifer C, Talwar P, Gudeloglu A, Mahmoud AMA, Terras K, Yazbeck C, Nebojsa B, Durairajanayagam D, Mounir A, Kahn LG, Baskaran S, Pai RD, Paoli D, Leisegang K, Moein MR, Malik S, Yaman O, Samanta L, Bayane F, Jindal SK, Kendirci M, Altay B, Perovic D, Harlev A. Male Oxidative Stress Infertility (MOSI): Proposed Terminology and Clinical Practice Guidelines for Management of Idiopathic Male Infertility. World J Mens Health. 2019 Sep;37(3):296-312. doi: 10.5534/wjmh.190055. Epub 2019 May 28. PMID 31081299